CLINICAL TRIAL: NCT02918604
Title: Peripheral Veins Cannulation in Children Using Veinsite: a Randomized Clinical Trial
Brief Title: Pediatric Veins Cannulation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Emanuele Rossetti, MD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-INNCB 11-2013
Record Dates: First submitted 2016-09-20; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Successful Vein Cannulation at First Attempt
Keywords: peripheral vein access; infrared; pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B : veinsite access (Other): infrared technology vein access
  Interventions: Device: infrared technology: Veinsite
- A: control group (Active Comparator): conventional vein access
  Interventions: Device: infrared technology: Veinsite

INTERVENTIONS:
Device: infrared technology: Veinsite — peripheral vein access performed with Veinsite support by expert paediatric anaesthesiologists and intensivists

SUMMARY:
multicenter, prospective and cohort study to evaluate infrared technology for identifying and and indwelling peripheral veins in 0 up to 4 years old children.

DETAILED DESCRIPTION:
AIM OF THE STUDY The primary objective of this study is to determine the success rate at first attempt of peripheral veins cannulation in small children (<5yrs) and infants (<1yr) of Veinsite compared with traditional palpation method performed by skilled operators.

The secondary objective of this study is to determine the time to cannulation using the two techniques, the difference in visualized veins using the Veinsite or the direct visualization and palpation of the patients' skin, cannula indwelling time and complications related to the procedure.

DESIGN Prospective randomized controlled study

Population

It is expected to recruit 60 pediatric patients undergoing peripheral vein cannulation with known difficulties according the difficult venous access score (DIVA) (6) in the following centers:

1. Fondazione IRCCS Istituto Neurologico "C.Besta" , Milano
2. Ospedale Pediatrico Bambino Gesù, IRCCS, Roma

Duration of study Patient will be followed from the day of peripheral vein cannulation till the peripheral cannula will be removed (max 3 days) in order to assess any cause of venous extravasation. The recruitment phase is supposed to be 6 months after achieving the ethical-administrative authorization.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female children from 1 month to 5 years Of age
* American Society of Anesthesiologists Classification (ASA) I: without systemic disease
* American Society of Anesthesiologists Classification (ASA) II: moderate systemic disease
* American Society of Anesthesiologists Classification (ASA) III: severe systemic disease that limits normal activity, without invalidity.
* Scheduled for any indication of peripheral venous line placement
* Admission to an Intensive Care Unit, Neurosurgery ward or pediatric ward of one of the hospitals included
* Children whose parents (or legal tutors) have given their informed written consent

Exclusion Criteria:

* Any contraindication for peripheral line placement
* Children whose parents (or legal tutors) denied their own consensus

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
success of peripheral vein access positioning | 2 year
  to determine the success rate at first attempt of peripheral veins cannulation in small children (<5yrs) and infants (<1yr) of Veinsite compared with traditional palpation method performed by skilled operators.

SECONDARY OUTCOMES:
impact of DIVA score(difficult vein access score) on time of success number of participants with treatment-related peripheral vein cannulation failure | 2 year
  of this study is to determine the time to cannulation using the two techniques, the difference in visualized veins using the Veinsite or the direct visualization and palpation of the patients' skin, cannula indwelling time and complications related to the procedure.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reigart JR, Chamberlain KH, Eldridge D, O'Brien ES, Freeland KD, Larsen P, Goff D, Hartzog TH. Peripheral intravenous access in pediatric inpatients. Clin Pediatr (Phila). 2012 May;51(5):468-72. doi: 10.1177/0009922811435164. Epub 2012 Jan 20. PMID 22267855
- [Background] Chapman LL, Sullivan B, Pacheco AL, Draleau CP, Becker BM. VeinViewer-assisted Intravenous catheter placement in a pediatric emergency department. Acad Emerg Med. 2011 Sep;18(9):966-71. doi: 10.1111/j.1553-2712.2011.01155.x. Epub 2011 Aug 19. PMID 21854488
- [Background] Kim MJ, Park JM, Rhee N, Je SM, Hong SH, Lee YM, Chung SP, Kim SH. Efficacy of VeinViewer in pediatric peripheral intravenous access: a randomized controlled trial. Eur J Pediatr. 2012 Jul;171(7):1121-5. doi: 10.1007/s00431-012-1713-9. Epub 2012 Mar 14. PMID 22415409
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490